CLINICAL TRIAL: NCT03172234
Title: Oral Amantadine Versus Gabapentin to Attenuate the Hemodynamic Response to Laryngoscopy and Tracheal Intubation and Their Effect on β-endorphin
Brief Title: Oral Amantadine Versus Gabapentin to Attenuate the Response to Laryngoscopy and Tracheal Intubation
Acronym: 15/5/2017
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ghada Mohammed AboelFadl (Other)
Responsible Party: Sponsor-Investigator, Ghada Mohammed AboelFadl, principal-investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Assuit universty
Record Dates: First submitted 2017-05-20; First posted 2017-06-01 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Effect of Laryngoscopy and Tracheal Intubation
Keywords: β-endorphins,laryngoscopy and tracheal intubation
MeSH Terms: interventions — Amantadine; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- amantadine group (Group A) (Active Comparator): the patients will receive oral amantadine sulfate using the dose 100 mg 120 minutes prior to the surgery, 5 ml saline IV 5 minutes before intubation.
  Interventions: Other: oral amantadine sulfate
- gabapentin group(Group B) (Active Comparator): the patients will receive oral gabapentin using the dose 800 mg 120 minutes prior to surgery,5 ml saline IV 5 minutes before intubation.
  Interventions: Drug: oral gabapentin
- control group (group C) (Placebo Comparator): the patients will receive placebo oral tablet 120 minutes prior to surgery, IV fentanyl 2µ/kg in 5 ml saline 5 minutes before intubation.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Other: oral amantadine sulfate — In amantadine group:the patients will receive100 mg oral amantadine sulfate 90 minute prior to the surgery
  Other Names: infex
  Arms: amantadine group (Group A)
Drug: oral gabapentin — In gabapentin group: the patients will receive oral 800 mg gabapentin 90 minute prior to the surgery
  Other Names: gabapentin
  Arms: gabapentin group(Group B)
Drug: Placebo Oral Tablet — in control group : the patients will receive Placebo Oral Tablet 90 minute prior to the surgery
  Arms: control group (group C)

SUMMARY:
To evaluate the effect of oral amantadine versus gabapentin premedication on the hemodynamic response to laryngoscopy and tracheal intubation and their effect on β-endorphins.

DETAILED DESCRIPTION:
Direct laryngoscopy and passage of endotracheal tube through the larynx is a noxious stimulus, which can provoke untoward response in the cardiovascular, respiratory and other physiological systems. Gabapentin, is 1-aminomethyl cyclohexane acetic acid.Gabapentin is structurally related to the neurotransmitter gamma-aminobutyric acid (GABA). Gabapentin act in central nervous system CNS), it acts by decreasing the synthesis of neurotransmitter glutamate and by binding to the alpha 2 delta subunits of voltage dependent calcium channels.

Amantadine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist, and compared to ketamine, it is well tolerated with fewer side effects (mainly dizziness, sedation, and dry mouth). Amantadine's formulation permits the oral route for drug delivery, as well as the IV route. The side-effects profile of amantadine via all routes seems not to be harmful in appropriate dosages.. Amantadine has been clinically used as an antiviral drug, for dementia, and in the treatment of Parkinson's disease and spasticity. It is a non-competitive NMDA receptor antagonist, and compared to ketamine, it is well tolerated with fewer side effects (mainly dizziness, sedation, and dry mouth). Amantadine's formulation permits the oral route for drug delivery, as well as the IV route. The side-effects profile of amantadine via all routes seems not to be harmful in appropriate dosages.

In the central nervous system, beta-endorphins bind mu-opioid receptors and exert their primary action at presynaptic nerve terminals. However, instead of inhibiting substance P, they exert their analgesic effect by inhibiting the release of GABA, an inhibitory neurotransmitter, resulting in excess production of dopamine.

The investigators designed this study to prove the efficacy of oral amantadine versus gabapentin premedication on the hemodynamic response to laryngoscopy and tracheal intubation and their effect on β-endorphins.

ELIGIBILITY:
Inclusion Criteria:

* ASA I&II scheduled for elective spine surgery

Exclusion Criteria:

* Patient refusal
* Patients with ASA score III (with chronic kidney, lungs, Gastrointestinal tract, liver, or cardiovascular diseases)
* Pregnant or breastfeeding women.
* Allergy to any of the study medications and taking medications that could significantly interact with amantadine (tramadol, atropine, antipsychotic medications)
* diabetes mellitus, thyroid disease any endocrine disease
* Suspected difficult intubation or intubation time more than 30 second.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
effect of oral amantadine versus gabapentin premedication on laryngoscopy and tracheal intubation on β-endorphins. | baseline blood sample taken before drug administration and after 15 minutes after intubation and before skin incision
  analysis of change of β-endorphins in blood sample

SECONDARY OUTCOMES:
effect of oral amantadine versus gabapentin premedication on the Mean arterial blood pressure due to laryngoscopy and tracheal intubation | baselineMAP before drug administration and after 15 minutes after intubation and before skin incision
  change of Mean arterial blood pressure
effect of oral amantadine versus gabapentin premedication on the heart rate due to laryngoscopy and tracheal intubation | baseline heart rate before drug administration and after 15 minutes after intubation and before skin incision
  change of heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Abualauon Elpiplaoy, MD, Principal Investigator — Assiut University; Ahmed El shanawany, MD, Study Chair — Assiut University; Azza Abo Elfadl El Sayed, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No